CLINICAL TRIAL: NCT06929052
Title: An Open Label, Randomized, Balanced, Two-treatment, Single Period, Parallel, Single Dose, Subcutaneous Administration, Comparative Pharmacokinetic Study of ADL-018 Injection 150 mg/mL Solution in a Single Dose Pre-filled Autoinjector Compared to ADL-018 Injection 150mg/mL Solution in a Single Dose Pre-filled Syringe in Normal, Healthy, Adult Subjects Under Fasting Conditions
Brief Title: An Open Label, Randomized, Parallel, Comparative Pharmacokinetic Study in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kashiv BioSciences, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADL-018 Autoinjector
Record Dates: First submitted 2025-01-31; First posted 2025-04-15 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Healthy Adult Subjects
Keywords: Xolair

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- test product (Experimental): Test product (A): ADL-018 Injection 150 mg/mL solution in a single dose pre-filled autoinjector manufactured/supplied by Kashiv BioSciences LLC, USA.
  Interventions: Device: ADL-018 Autoinjector
- reference product (Active Comparator): Reference Product (B): ADL-018 Injection 150mg/mL solution in a single dose pre-filled syringe manufactured/supplied by Kashiv Biosciences LLC, USA
  Interventions: Drug: ADL-018 Injection

INTERVENTIONS:
Device: ADL-018 Autoinjector — Test product (A): ADL-018 Injection 150 mg/mL solution in a single dose pre-filled autoinjector manufactured/supplied by Kashiv BioSciences LLC, USA.
  Arms: test product
Drug: ADL-018 Injection — Reference Product (B): ADL-018 Injection 150mg/mL solution in a single dose pre-filled syringe manufactured/supplied by Kashiv BioSciences LLC, USA
  Arms: reference product

SUMMARY:
The Goal of these study is to assess the comparative pharmacokinetics of Test Product (A): ADL-018 Injection 150 mg/mL solution in a single dose pre-filled autoinjector, manufactured by Kashiv Biosciences LLC, USA with Reference Product (B): ADL-018 Injection 150mg/mL solution in a single dose pre-filled syringe manufactured by Kashiv Biosciences LLC, USA in healthy, adult human subjects. and also to assess safety and tolerability of investigational product.

DETAILED DESCRIPTION:
An Open label, Randomized, Balanced, Two-treatment, Single Period, Parallel, Single dose, Subcutaneous administration, comparative pharmacokinetic study of ADL-018 Injection 150 mg/mL solution in a single dose pre-filled autoinjector compared to ADL-018 Injection 150mg/mL solution in a single dose pre-filled syringe in normal, healthy, adult subjects under fasting conditions.

The total expected study duration of the clinical part is approximately 127 days from the day of check-in to end study visit.

Approximate volume of blood loss in the study will be 150 mL.

Handling of Pharmacokinetic Samples After collection, blood samples will be allowed to clot at room temperature for at least 30 to 60 minutes and then will be placed in a refrigerated centrifuge, and then spun at 3000 rpm (± 50 rpm) under refrigeration at 4° C (±2° C) for 10 minutes. The serum will be divided into two aliquots in such a way that the Aliquots#01 (primary aliquot) will contain at least 1.2 mL of serum and the remaining quantity of serum will be transferred into the Aliquots#02 (secondary aliquot) and will be stored in freezer at -70ºC ± 10ºC at the clinical facility until shipment to the analytical facility.

The time between the end of centrifugation and placement of samples in the Freezer shall not exceed 45 minutes (+ 15 minutes).

The samples will be stored in a freezer at -70ºC ± 10ºC at the analytical facility until analyzed (all the temperature excursions will be handled as per in-house SOP).

In case of any processing error due to any reason (e.g. mixing of sample while segregation, mechanical failure in centrifuge, etc.) during the sample processing, re-spun the sample (s) under the same conditions, if required.

Note:

Transfer of serum samples into the freezer shall take place as soon as possible so the total elapsed time from blood collection to placement of serum samples in the freezer does not exceed 120 minutes.

Statistical analyses will be performed on ln-transformed pharmacokinetic parameters Cmax, AUC0-t and AUC0-inf for Omalizumab using the SAS® software version 9.4 or higher. The pharmacokinetic analysis will include evaluable data from all the subjects who comply with the protocol sufficiently, complete the study and for whom the PK profile can be adequately characterized. The ln-transformed pharmacokinetic parameters e.g. Cmax, AUC0-t and AUC0-∞ will be analyzed using a PROC MIXED effect ANOVA model with the main effect of treatment as fixed effect. A separate ANOVA model will be used to analyze each of the pharmacokinetic parameters. Treatment effects will be tested at the 0.05 level of significance against the residual error (mean square error or MSE) from the ANOVA as the error term. The power of ANOVA test to detect a 20% mean difference between test and reference formulations will be reported. Difference of LSMs will be calculated for ln-transformed pharmacokinetic parameters Cmax, AUC0-t and AUC0-∞. The difference will be of the form: Test Product (A) - Reference Product (B). Ratios of means will be expressed in percentage by taking the anti-ln value of difference of LSM. The geometric mean values will be reported. 90% confidence intervals for the difference between investigational product LSMs will be calculated for the pharmacokinetic parameters Cmax, AUC0-t and AUC0-∞ using ln-transformed data. The confidence intervals will be expressed as a percentage relative to the LSM of the reference product.

Based on the 90% confidence intervals for the difference of means of lntransformed Pharmacokinetic Parameters Cmax, AUC0-t and AUC0-∞ conclusions will be drawn whether the test product is bioequivalent to the reference product.

under fasting condition. The acceptance range for bioequivalence is 80.00-125.00% for the 90% confidence intervals for the difference of means of ln-transformed Cmax, AUC0-t and AUC0-∞ with respect to Omalizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 65 years of age, inclusive, at the time of dosing.
2. Subject should be having serum total IgE ≤ 100 IU/ml at the time of screening
3. Gender: Male and/or non-pregnant, non-lactating female. Female of childbearing potential must have a negative serum pregnancy test performed within 28 days prior to dosing day.
4. Male subjects and/or female subject's partner must agree to use acceptable form of contraception which includes vasectomy, or use condoms, or spermicide in addition to female contraception for additional protection against conception from screening until 156 days after administration of the study medication.
5. For female of childbearing potential, must agree to use acceptable forms of contraception from screening until 156 days after administration of the

   Investigational Product include the following:

   Non hormonal intrauterine device in place, or Barrier methods containing or used in conjunction with a spermicidal agent, or Surgical sterilization or Practicing sexual abstinence.

   Female will not be considered of childbearing potential if one of the following is reported and documented on the medical history:

   Postmenopausal with spontaneous amenorrhea for at least one year, or Spontaneous amenorrhea for more than 6 months and less than one year with Serum Follicular Stimulating Hormone (FSH) level > 40 IU/L, or Bilateral oophorectomy with or without a hysterectomy and an absence of bleeding for at least 6 months, or Total hysterectomy and an absence of bleeding for at least 3 months.
6. BMI: 18.5 to 32.0 kg/m2, both inclusive; BMI value should be rounded off to one significant digit after decimal point (e.g., 32.04 rounds down to 32.0, while 18.49 rounds up to 18.5).
7. Volunteers having body weight ≥50.0 kg or ≤ 90.0 kg.
8. Able to communicate effectively with study personnel.
9. Willing to provide written informed consent to participate in the study.
10. Non-smokers and non-tobacco users (i.e., having no past history of smoking and tobacco consuming for at least one year prior to study).
11. All volunteers must be judged by the principal and /or sub investigator principal or sub-investigator or physician as normal and healthy during a pre-study safety assessment performed within 28 days of the study medication administration which will include:

A comprehensive physical examination, medical history, vital sign assessments, 12-lead electrocardiogram (ECG) with no clinically significant finding.

Exclusion Criteria:

1. History of allergic responses to study drug or other related drugs, or any of its formulation ingredients.
2. History of allergic reactions or sensitivity to latex or latex derived products.
3. Have significant diseases or clinically significant abnormal findings during screening [medical history, comprehensive physical examination, vital signs, laboratory evaluations and ECG].
4. Any disease or condition like diabetes, psychosis or others, which might compromise the hemopoietic, gastrointestinal, renal, hepatic, cardiovascular, respiratory, central nervous system or any other body system.
5. History of helminthic or parasitic infection.
6. History of immunological disorders or presence of bronchial asthma.
7. Use of any hormone replacement therapy within 3 months prior to the study medication administration.
8. Use of any depot injection or implant of any drug within 3 months prior to the study medication administration.
9. Use of CYP enzyme inhibitors or inducers or St. John's Wort within 30 days prior to the study medication administration (see https://druginteractions. medicine.iu.edu/MainTable.aspx).
10. Reports a history of drug or alcohol addiction or abuse within the past 1 year.
11. History or evidence of drug dependence.
12. History of difficulty with donating blood or difficulty in accessibility of veins.
13. A positive hepatitis screen (hepatitis B surface antigen, hepatitis C antibody).
14. A positive test result for HIV antibody.
15. Demonstrates a positive drug screen, cotinine, or alcohol test during screening
16. Volunteers who have received any investigational drug/product within 30 days prior to the study medication administration.
17. Volunteers who have donated blood or loss of blood between 101 mL to 499 mL within 30 days prior to dosing or a blood donation of more than 499 mL within 56 days prior to dosing for male volunteers and 84 days prior to dosing for female volunteers.
18. Intolerance to venipuncture Demonstrates, in the opinion of the study staff, inadequate vein or vein unsuitable for repeated venipuncture (e.g. vein difficult to locate, access or puncture, vein with a tendency to rupture during or after puncture).

20) Any food allergy, intolerance, restriction or special diet that, in the opinion of the principal investigator or sub-investigator, could contraindicate the volunteer's participation in this study. 21) If, in the opinion of the investigator, the subject is not suitable for the study.

22) Institutionalized volunteers. 23) Use of any prescribed medications and/or Monoamine Oxidase Inhibitor (MAOI) within 14 days prior to the study medication administration. 24) Use of any herbal or dietary supplements or over-the-counter medications (Tylenol, Advil, etc.) or therapeutic dose of vitamins (including vitamin water) products, etc., within 7 days prior to the study medication administration. 25) Use of any products containing Seville oranges, grapefruit and pomelo within 7 days prior to the study medication administration.

26) Use of any products containing broccoli, brussels sprouts, and char-grilled meat within 14 days prior to the study medication administration.

27) Ingestion of any caffeine/xanthine containing products (coffee, tea, soft drinks, chocolate, energy drinks, etc.), alcohol and/or other alcohol containing products, foods containing poppy seeds within 48 hours prior to the study medication administration. 28) Ingestion of any beverages containing more than 5% fruit juice (fruit drinks, fruit punches, fruit cocktails, fruit , or other products containing 5% or less of fruit juice will be allowed) within 48 hours prior to the study medication administration. 29) Ingestion of any unusual diet, for whatever reason (e.g.: low sodium) for three weeks prior to the study medication administration.

30) History of anaphylactic shock. 31) History of being on allergy vaccine therapy. 32) Intravenous (IV) immunoglobulin G (IVIG), or plasmapheresis within 90 days prior to the study medication administration.

Subjects with current malignancy, history of malignancy, or currently under work-up for suspected malignancy except non-melanoma skin cancer that has been treated or excised and is considered resolved. 34) Female volunteer who has used implanted or injected hormonal contraceptives anytime during the 6 months prior to study or used hormonal contraceptives within 3 months before dosing.

35) Pregnant, breastfeeding, or intends to become pregnant over the course of the study.

36) Difficulty in fasting or consuming standardized meals. 37) Reports a clinically significant illness during the 28 days prior to dosing (as determined by the investigator and/or designee). 38) Reports undergoing any kind of surgical procedures with general anesthesia within 3 months prior to dosing.

39) Presence of tattoos or other skin conditions on both the left and right upper outer arms at the injection site based on PI discretion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2025-01-29 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter | Baseline to day 126
  Cmax
Pharmacokinetic parameter | Baseline to day 126
  AUC0-t
Pharmacokinetic parameter | baseline to day 126
  AUC0-inf

CONTACTS AND LOCATIONS:
Locations (1):
- Cliantha Research, Mississauga, ON L4W 1A4, Canada